CLINICAL TRIAL: NCT04127201
Title: En_Línea. An Online Treatment to Change Lifestyle in Overweight and Obesity: Study Protocol for a Randomized Controlled Trial
Brief Title: En_Línea. An Online Treatment to Change Lifestyle in Overweight and Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Carmina Saldaña, PhD, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00003099
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Overweight; Obesity
Keywords: "online therapy"; "weight loss control program"; Internet
MeSH Terms: conditions — Overweight; Obesity | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online intervention, en_línea (Experimental): Participants will be provided with a username and a password to acess to a website. en_línea program is an online adaptation of the LEARN program. The five treatment areas are: Lifestyle, Exercise, Attitudes, Relationships and Nutrition. We have designed and developed a website (www.programaenlinea.org) with 17 weekly treatment sessions and an exclusive mobile application for self-recording.
  Interventions: Behavioral: en_línea
- Standard group therapy (Active Comparator): Participants in this arm will received a 10 sessions of standard primary care group therapy. Sessions 1 and 2 will be weekly and sessions from 3 to 10 will be biweekly. Sessions, between 8 and 10 participants, will be conducted by a specialized psychologist and they will last 90 minutes. Treatment areas will be the same as en_línea, beginning with nutrition and exercise and a progressive incorporation of the other topics. Material to work at home and self-recording will be provided in paper.
  Interventions: Behavioral: Group therapy
- Control group (No Intervention): Participants in the control group only will receive a biweekly newsletter by email without feedback. They will be provided with material and instructions to self-record their daily meals and exercise. The newsletter only will content basic information about nutrition and exercise.

INTERVENTIONS:
Behavioral: en_línea — This is an online adaptation of the LEARN program. A self-help weight control program developed by Kelly Brownell in 2004.
  Other Names: Web-based weight control program
  Arms: Online intervention, en_línea
Behavioral: Group therapy — This is a traditional behavioral weight control program
  Arms: Standard group therapy

SUMMARY:
A randomized controlled trial to test the effectiveness of an online weight control program, called en_línea, comparing with a standard group therapy and a control group

DETAILED DESCRIPTION:
This is a randomized controlled trial with three intervention arms: en_línea, standard group therapy and control group. To perform this study, 305 adults (18-65 years) with overweight type II (27-29.9 kg/m2) or obesity type I (30-34.9 kg/m2) will be invited to participate. Interventions will last 17 weeks with follow-ups 1, 3, 6 and 12 months after the post-treatment appointment. The primary outcome will be post-treatment weight loss and the maintenance during the follow-ups. Secondary outcomes will be adherence rates, drop outs and quality of life. Participants will be assessed before randomization and they will be sign an inform consent.

ELIGIBILITY:
Inclusion Criteria:

1. Overweight type II or obesity type I. BMI between 27 and 34.9 kg/m2
2. Age between 18 and 65 years old
3. Compliance with all evaluation phases.

Exclusion Criteria:

1. Presence of several physical disease, i.e. diabetes, hypertension, cancer or metabolic disorders
2. Presence of several psychological problem, i.e. depression, anxiety
3. Presence of other eating disorders, i.e. anorexia nervosa, bulimia nervosa, binge eating disorders
4. Use of drugs, i.e. slimming, anovulatory or psychotropic
5. Pregnancy or planned pregnancy for the next six months
6. Following another weight control program at the time of selection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 4 months
  5%-10% of weight loss respect the initial weight
Maintenance of weight loss 1 month follow-up | 1 month follow-up
  Maintenance of weight loss
Maintenance of weight loss 3 months follow-up | 3 months follow-up
  Maintenance of weight loss
Maintenance of weight loss 6 months follow-up | 6 months follow-up
  Maintenance of weight loss
Maintenance of weight loss 12 months follow-up | 12 months follow-up
  Maintenance of weight loss

SECONDARY OUTCOMES:
Adherence | 4 months
  80% of completed website activities and 80% of self-records
Drop out | 4 months
  Percentage of participants who finish the treatment
Quality of life test measures | 4 months
  Questionnaire of Quality of Life provided by the LEARN program

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Terapia de Conducta, University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Research team have to meet and make a decision about this field

REFERENCES:
- [Derived] Varela C, Saldana C. En_Linea. An online treatment to change lifestyle in overweight and obesity: study protocol for a randomized controlled trial. BMC Public Health. 2019 Nov 21;19(1):1552. doi: 10.1186/s12889-019-7928-1. PMID 31752815